CLINICAL TRIAL: NCT04233203
Title: Effectiveness and Safety of Insulin Faster Aspart on Continuous Subcutaneous Insulin Infusion Treated Adult Type 1 Diabetes Mellitus Patients in Routine Clinical Practice
Brief Title: Faster Aspart on Insulin-pump Treated T1DM Patients
Acronym: realFACI
Status: Completed | Type: Observational
Sponsor: Jesús Moreno Fernández (Other)
Collaborators: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor-Investigator, Jesús Moreno Fernández, Endocrinology and Nutrition Service, MD, PhD Affiliation: Castilla-La Mancha Health Service, Castilla-La Mancha Health Service
Organization: Castilla-La Mancha Health Service (Other)
Other Study IDs: C-302
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Type 1 Diabetes
Keywords: insulin pump; Faster aspart; insulin; glycemic variability
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Insulin Aspart; Insulin Infusion Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Faster Aspart: All T1DM adult patients attended in Ciudad Real General University Hospital and treated with CSII and insulin Faster Aspart.
  Interventions: Drug: Insulin Faster Aspart; Device: Insulin pump

INTERVENTIONS:
Drug: Insulin Faster Aspart — Currently receiving Faster Aspart during 3 or more months.
  Other Names: Fiasp
Device: Insulin pump — Currently receiving CSII therapy during 6 or more months.
  Other Names: Medtronic 640G; Medtronic 670G; T Slim X2; Accucheck Insight

SUMMARY:
Observational retrospective study about effectiveness and safety of insulin Faster Aspart on continuous subcutaneous insulin infusion treated adult Type 1 Diabetes Mellitus (T1DM) patients in routine clinical practice.

DETAILED DESCRIPTION:
Cross-sectional retrospective analysis about effectiveness and safety of insulin Faster Aspart on continuous subcutaneous insulin infusion treated adult Type 1 Diabetes Mellitus (T1DM) patients in routine clinical practice.

All clinical variables are gathered from two EMR softwares (Mambrino XXI and Carelink Pro®).

Data analysis is conducted using SPSS (Chicago, IL) statistics software. Results are presented as mean ± SD values or percentages. A paired Student's t-test or a Wilcoxon signed-rank test were used for the analysis of differences. Comparisons between proportions were analyzed using a chi-squared test. A P value < 0.05 was considered statistically significant.

The protocol was approved by the reference Castilla-La Mancha Public Health Institute Ethic Committee. All participants provided written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age.
* Diagnosed of Type 1 Diabetes Mellitus.
* Be attended in Ciudad Real General University Hospital.
* Current treated with CSII (CSII cohort) during ≥6 months.
* Current treated with insulin Faster Aspart during ≥3 months.

Exclusion Criteria:

* Less than 18 years old.
* Other types of diabetes mellitus.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years of age) T1DM patients on CSII with Faster Aspart attended to care in our consults were eligible.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
MAGE | 3 months
  Differences from basal to 3 months after Faster Aspart initiation on Mean Amplitude of Glucose Excursions (MAGE).

SECONDARY OUTCOMES:
VCo | 3 months
  Differences from basal to 3 months after Faster Aspart initiation Variation Coefficient (VCo).
M100 | 3 months
  Differences from basal to 3 months after Faster Aspart initiation on M100.
GRADE | 3 months
  Differences from basal to 3 months after Faster Aspart initiation on Glycemia Risk Assessment Diabetes Equation (GRADE).
J-index | 3 months
  Differences from basal to 3 months after Faster Aspart initiation on J-index.
MODD | 3 months
  Differences from basal to 3 months after Faster Aspart initiation on MODD.
CONGA | 3 months
  Differences from basal to 3 months after Faster Aspart initiation on CONGA.
HbA1c | 3 months
  Differences from basal to 3 months after Faster Aspart initiation on Hemoglobin A1C (HbA1C).
Hypoglycemic frequency | 3 months
  Differences from basal to 3 months after Faster Aspart initiation on hypoglycemic frequency.
TIR-TAR-TUR | 3 months
  9. Differences from basal to 3 months after Faster Aspart initiation on time in range, time above range and time under range.

OTHER OUTCOMES:
Other glycemic outcomes | 3 months
  Other glycemic control differences from basal to 3 months after Faster Aspart initiation: capillary blood glucose, interstitial blood glucose, self-monitoring of blood glucose (SMBG) daily frequency, severe hypoglycemia frequency.
Weigh | 3 months
  Differences from basal to 3 months after Faster Aspart initiation on weight
Insulin dose | 3 months
  Daily insulin doses (basal and bolus) and bolus insulin daily frequency.
Local adverse effects | 3 months
  Faster Aspart related local adverse effects: itchiness, stinginess, pain, erythema, weal.
Catheters problems | 3 months
  Incidences on insulin-pump catheters: obstructions, deformations.
Catheter change frequency | 3 months
  Insulin-pump catheter change frequency
Severe adverse effects | 3 months
  Faster Aspart severe adverse effects: ketosis, diabetic ketoacidosis, death.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Alberto Garcia Seco, RN, Study Chair — Ciudad Real General University Hospital
Locations (1):
- Obispo Rafael Torija, St., Ciudad Real, Spain

REFERENCES:
- [Derived] Moreno-Fernandez J, Garcia-Seco JA, Virlaboa-Cebrian R, Seco AM, Munoz-Rodriguez JR, Gomez-Romero FJ. Faster-acting insulin aspart reduces glycaemic variability in sensor-augmented pump treated type 1 diabetes patients. Endocrinol Diabetes Nutr (Engl Ed). 2023 Jun-Jul;70(6):389-395. doi: 10.1016/j.endien.2021.12.012. PMID 37356876